CLINICAL TRIAL: NCT00442234
Title: Pharmacokinetic/Pharmacodynamic Study of Monteplase ("Cleactor") in Acute Pulmonary Embolism
Brief Title: Post-marketing Study of Monteplase ("Cleactor") in Patients With Acute Pulmonary Embolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E6010-J081-591
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2010-01

CONDITIONS: Pulmonary Embolism
Keywords: Acute; pulmonary; embolism; accompanying; hemodynamic; instability
MeSH Terms: conditions — Pulmonary Embolism; Embolism | interventions — monteplase

INTERVENTIONS:
Drug: Monteplase

SUMMARY:
To investigate PK and coagulating and fibrinolytic parameter profiles (PD) at the approved dose (13,750 - 27,500 IU/kg) in patients with acute pulmonary embolism accompanying hemodynamic instability.

ELIGIBILITY:
Inclusion Criteria:

1) Patients who consent for study participation and submit written informed consent with free will by patient or legally authorized representative.

2) Patients aged between 20 years or above and under 75 years old at the time of obtaining informed consent.

3) Patients with acute pulmonary embolism within 5 days after the onset.

4) Patients with acute pulmonary embolism with hemodynamic instability and fulfill all of the following 4 items:

1. Confirmed to have thrombi, emboli, or disorders in pulmonary circulation detected by pulmonary angiography or computed tomography.
2. Confirmed to have any of the following right ventricular overloads by echocardiography:

   i) Dilation of right ventricular cavity or hypokinesis in ventricular wall

   ii) Floating thrombi in pulmonary artery and right heart

   iii) Paradoxical motion in the interventricular septum

   iv) Disparity of tricuspid regurgitation pressure

   v) Enlargement of pulmonary artery
3. Mean pulmonary arterial pressure (PAP) is 20 mmHg or above
4. PaO2 is 65 mmHg or below (confirmed by blood gas analysis)

Exclusion Criteria:

1. Patients with concurrent hemorrhage (e.g., gastrointestinal bleeding, urinary tract bleeding, retroperitoneal bleeding, intracranial bleeding, or hemoptysis).
2. Patients who underwent intracranial or spinal operation or injury within 2 months prior to study treatment.
3. Patients with intracranial tumor, arteriovenous malformation, or aneurysm
4. Patients with hemorrhagic diathesis (e.g., vascular purpura, thrombocytopenia, hemophilia)
5. Patients with hypertension of systolic blood pressure >=180 mmHg or diastolic pressure >= 110 mmHg.
6. Patients with a history of cerebrovascular disorder (e.g., cerebral infarction, intracerebral hemorrhage).
7. Patients with severe hepatic disorder (e.g., cirrhosis, severe hepatitis) or severe renal disorder (e.g., renal failure).
8. Patients received thrombolytic drug (t-PA or urokinase) within 7 days prior to study treatment.
9. Patients with pulmonary cardiac arrest (CPA).
10. Patients with a history of hypersensitivity to monteplase or protein preparations.
11. Pregnant women, women suspected of being pregnant, women who desire to become pregnant during a period between obtaining informed consent to the final observation, or lactating women.
12. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

PRIMARY OUTCOMES:
Monteplase antigen levels in plasma; Monteplase activity in plasma; parameters of coagulating and fibrinolytic system (Plasminogen activity, a2-PI, PIC, fibrinogen, D-dimer).

SECONDARY OUTCOMES:
Symptoms and signs of acute pulmonary embolism; pulmonary thrombosis; echocardiography; pulmonary arterial pressure; blood gas; vital signs; laboratory tests (e.g., hematology and blood chemistry); adverse events; concomitant therapies; dosing regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Musha, Study Director — Department Marketed Product Research, Clinical Research Center
Locations (2):
- Japan (2):
  - Yokohama, Kanagawa
  - Bunkyo-ku, Tokyo